CLINICAL TRIAL: NCT06560099
Title: Standard Oxytocin Versus High Dose Oxytocin to Control Postpartum Hemorrhage in High Risk Pregnancy During Elective Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Laura 1 protocol
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (standard oxytocin dose) (Active Comparator)
  Interventions: Drug: Oxytocin
- Group B (high dose oxytocin) (Active Comparator)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — will receive 10 IU oxytocin intravenous bolus over one min and infusion of 10 IU oxytocin in 500 ml of 0.9 saline over four hours.

SUMMARY:
Controlling hemorrhage during and after a cesarean section reduces significantly maternal mortality and morbidity and the present study is important for detection of the effectiveness of routinely increasing the oxytocin dose instead of using the standard dose only in preventing postpartum hemorrhage and additional use of uterotonics in the first 24 hours after cesarean section for high risk pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* - Medical disorders ie: Hypertensive diseases with pregnancy - Diabetes Mellitus - Collagen diseases - Coagulopathies - Cardiac diseases - Anemia
* History of postpartum hemorrhage
* Placental disorders ie: placenta previa
* Infertility and ICSI
* High Parity
* History of Endometriosis
* Fetal disorders (IUGR, IUFD, Preterm, Congenital anomalies, oligohydramnios or polyhydramnios, macrosomia)
* Preterm labor on uterine relaxants
* Twins pregnancy
* Patients on antiplatelets and anticoagulants
* Uneventful antenatal care

Exclusion Criteria:

* - Oxytocin Allergy
* Normal uncomplicated pregnancy
* Emergency cesarean section
* Exhausted uterus due to trial of normal labor
* Couvelaire uterus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
blood loss | at the end of the operation
  measure blood in suction, towels and pads

SECONDARY OUTCOMES:
haemoglobin | immediate preoperative
  by laboratory asessment
haemoglobin | 6 hours postoperative
  by laboratory asessment

IPD SHARING:
Plan to Share IPD: No